CLINICAL TRIAL: NCT01752738
Title: The Influence of Chronic Kidney Disease on Intestinal Transport of Gut Microbial Metabolites
Brief Title: Intestinal Transport of Microbial Metabolites in Chronic Kidney Disease
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S54909
Record Dates: First submitted 2012-12-11; First posted 2012-12-19 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma, urine, faeces
Oversight: Data Monitoring Committee: No

SUMMARY:
Chronic kidney disease is associated with the accumulation of various metabolites, i.e., uremic retention solutes. Evidence is mounting that the colonic microbiome contributes substantially to these uremic retention solutes. Indoxyl sulfate and p-cresyl sulfate are among the most extensively studied gut microbial metabolites, and are associated with cardiovascular disease, chronic kidney disease progression and overall mortality. Mechanisms governing their intestinal uptake and metabolism, however, are currently unknown. The investigators aim to explore these transport characteristics in depth. Therefore, colonic biopsies will be sampled of patients with chronic kidney disease, analyzed and compared to available data of healthy controls. Insights in the mechanisms controlling intestinal transport and metabolism of indoxyl sulfate and p-cresyl sulfate is certainly relevant as it might lead to novel therapeutic targets in the treatment of chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 85 years
* Chronic kidney disease ≤ stage III (KDOQI), i.e., estimated glomerular filtration rate (MDRD) < 60 ml/min/m² or need of dialysis therapy 27
* Scheduled colonoscopy for diagnostic purposes
* Written informed consent

Exclusion Criteria:

* History of gastro-intestinal disease (e.g., inflammatory bowel disease)
* History of colon surgery
* Recipient of a renal or other solid organ transplant
* Exposure to antibiotics or drug therapy with a known influence on intestinal transporters (e.g., P-gp) or enzymes during 2 weeks before colonoscopy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the nephrology outpatient clinic and dialysis center at University Hospital Leuven, Belgium.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2013-12; Primary Completion 2021-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage change in number of intestinal drug transporters and enzymes | 4 years
  Influence of chronic kidney disease on intestinal drug transporters and enzymes responsible for uptake and metabolism of microbial metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Bjorn Meijers, MD, PhD, Principal Investigator — UZ Leuven; Sander Dejongh, Principal Investigator — KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams Brabant, Belgium